CLINICAL TRIAL: NCT06791486
Title: Predicting Biological Age Using Electronic Health Records: An AI-Based Approach
Brief Title: AI-Driven Prediction of Biological Age With EHR
Status: Recruiting | Type: Observational
Sponsor: The Eye Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Kang Zhang, Chief Scientist, Wenzhou Medical University
Other Study IDs: Biological Age
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Biological Age
Keywords: Biological Age; electronic health records; AI prediction; aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Biologically Younger Group: Participants whose biological age is predicted to be younger than their chronological age.
  Interventions: Other: AI-assisted predictive model
- Biologically Older Group: Participants whose biological age is predicted to be older than their chronological age.
  Interventions: Other: AI-assisted predictive model

INTERVENTIONS:
Other: AI-assisted predictive model — This study utilizes an AI-assisted predictive model that analyzes multimodal data from electronic health records, including medical history, laboratory results, imaging data, and lifestyle factors, to estimate biological age. The model employs deep learning algorithms to predict biological age, compare it to chronological age, and identify early signs of age-related health risks. The intervention is not a direct treatment or procedure but aims to develop a tool for predicting biological age to help personalize care and improve long-term health outcomes.

SUMMARY:
This is a multi-center, retrospective clinical study designed to evaluate the application and effectiveness of an AI-assisted predictive model for predicting biological age using electronic health records (EHR). The study will analyze various health data points, including medical history, laboratory results, and clinical observations, to estimate the biological age of patients. By comparing biological age with chronological age, the study aims to assess the accuracy of the model and its potential in identifying age-related health risks and improving patient care.

DETAILED DESCRIPTION:
Biological age prediction is crucial for assessing overall health, determining the risk of age-related diseases, and providing personalized healthcare. While chronological age is a key factor, it does not always reflect an individual's true biological aging process. Early identification of accelerated biological aging and associated health risks can significantly impact early interventions and long-term health outcomes. In clinical practice, healthcare providers integrate a wide range of patient data, including medical history, laboratory test results, and clinical observations, to understand an individual's health status and predict potential future risks. As precision medicine becomes more important, the ability to predict biological age and personalize care plans is essential. Recent advancements in artificial intelligence and data analysis techniques have shown promise in enhancing the accuracy of biological age predictions. This study aims to develop an AI-assisted decision-making system by integrating multimodal data from electronic health records, laboratory results, clinical observations, and patient demographics. The objective is to improve diagnostic accuracy, optimize clinical workflows, and provide more personalized healthcare for patients by predicting biological age, identifying at-risk individuals, and improving health outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with comprehensive and accessible EHR data, including medical history, laboratory results, treatment data, imaging data (if available), and lifestyle factors (e.g., smoking, physical activity, diet).
2. Patients with no significant cognitive impairments that would prevent them from providing informed consent or participating in the study.
3. All participants must provide informed consent for the use of their medical data for research purposes.

Exclusion Criteria:

1. Patients with incomplete or missing critical EHR data such as medical history, laboratory results, or treatment data that are necessary for predicting biological age.
2. atients with severe cognitive disorders (e.g., dementia, significant mental disabilities) who are unable to provide informed consent or participate meaningfully in the study.
3. Patients with terminal illnesses or those with limited life expectancy where biological age predictions may not be relevant for the purposes of the study.

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of individuals who have received care at participating hospitals or healthcare centers with accessible electronic health records (EHR). Participants will include those with complete EHR data, including medical history, laboratory test results, imaging data, and lifestyle factors such as diet, physical activity, and smoking habits. The cohort will comprise both individuals who are healthy and those with chronic conditions or comorbidities to analyze biological age prediction across different health statuses. The study will be conducted across multiple healthcare facilities to ensure a diverse patient population representing a wide range of age groups, health conditions, and demographics.
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-04-02 (Estimated); Study Completion 2025-04-02 (Estimated)

PRIMARY OUTCOMES:
Biological Age Prediction Accuracy | 1 year
  The accuracy of the AI model in predicting biological age compared to chronological age. This will be evaluated using the Pearson Correlation Coefficient (PCC) to assess the strength of the correlation between predicted biological age and chronological age. Additionally, R-squared (R²) will be used to evaluate the proportion of variance in biological age explained by the model.

SECONDARY OUTCOMES:
Health Risk Correlation | 1 year
  The correlation between predicted biological age and various health risks, such as the development of chronic diseases (e.g., cardiovascular disease, diabetes), using PCC to evaluate the relationship between biological age predictions and health outcomes.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Nanfang Hospital, Guangzhou, Guangdong
  - First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The Eye Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No